CLINICAL TRIAL: NCT06803017
Title: The Effect of Music Intervention in Exercise and Sport on Problematic Smartphone Use, Psychopathological Symptoms, Self-Esteem, and Impulsivity Traits Among College Students in China
Brief Title: Music Intervention in Exercise and Sport on Problematic Smartphone Use, Psychopathological Symptoms Among College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: YALI ZHOU (Other)
Responsible Party: Sponsor-Investigator, YALI ZHOU, Principal Investigator, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YZHOU
Record Dates: First submitted 2025-01-17; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-10

CONDITIONS: Problematic Smartphone Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- combination of exercise and sport with fast-tempo music (Experimental)
  Interventions: Behavioral: combination of exercise and sport with fast-tempo music
- combination of exercise and sport with slow-temp music (Experimental)
  Interventions: Behavioral: combination of exercise and sport with slow-temp music
- combination of exercise and sport with no music (Experimental)
  Interventions: Behavioral: combination of exercise and sport with no music

INTERVENTIONS:
Behavioral: combination of exercise and sport with fast-tempo music — Fast-tempo music selected by the researcher with exercise training and sports training
  Arms: combination of exercise and sport with fast-tempo music
Behavioral: combination of exercise and sport with slow-temp music — Slow-tempo music selected by the researcher with exercise training and sports training
  Arms: combination of exercise and sport with slow-temp music
Behavioral: combination of exercise and sport with no music — Exercise training and sports training without music
  Arms: combination of exercise and sport with no music

SUMMARY:
This study is to examine the effect of music intervention in exercise and sport on problematic smartphone use, psychopathological symptoms, self-esteem, and impulsivity traits in smartphone users among Chinese college students. The aim is to compare the effects of the combination of exercise and sport with fast-tempo music, slow-tempo music, and no music.

ELIGIBILITY:
Inclusion Criteria:

* University students aged between 18 and 25 years old (male or female)
* No cognitive impairment and able to complete the questionnaire clearly

Exclusion Criteria:

* Students with recent injuries such as broken bones, congenital diseases such as heart disease, or other status conditions that prevent them from playing moderate-to-high-intensity sports
* Excluded students with mental diseases, physical disabilities, or those who were unable or unwilling to participate in the trial

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-10-07 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Smartphone Impact Scale (SIS) | 14 weeks
  The SIS is a 26-item scale developed in Italian to comprehensively account for smartphones' different cognitive, affective, social, and behavioural impacts in everyday life. The SIS dimensions were measured on a 5-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree).
Ryerson Social Anxiety Scales (RSAS) | 14 weeks
  The RSAS is a new self-report measure designed to assess the extent to which respondents experience fear or anxiety across several social situations (Situations scale), as well as the degree of distress and impairment associated with their social anxiety (Severity scale). Possible scores range from 0 to 28, with higher scores indicating higher social anxiety.
Impulsive Behavior Short Scale-8 (I-8) | 14 weeks
  The Impulsive Behavior Short Scale-8 (I-8) measures the psychological construct of impulsivity with four subscales comprising two items each (completion time < 1 min). I-8 consists of eight items measuring four personality facets that lead to impulsive behaviour: urgency, lack of premeditation, lack of perseverance, and sensation seeking. It was measured on a 4-point Likert scale, ranging from 1 (strongly agree) to 4 (strongly disagree).
Depression Anxiety Stress Scale 8-items (DASS-8) | 14 weeks
  The DASS-8 is an 8-item scale that evaluates stress, depression, and anxiety. Items are rated on a 4-point scale ranging from 0 (never or almost never) to 3 (almost always or always).
Multidimensional Self-Esteem Scale-12(MSES-12) | 14 weeks
  MSES-12 consists of six subscales comprising 12 items, each rated on a 7-point rating scale ranging from 1 (= not at all) to 7 (= very much) for items measuring the intensity and from 1 (= never) to 7 (= very much) for items measuring frequency.
The SCRAM (Sleep, Circadian Rhythms, and Mood) Questionnaire | 14 weeks
  The SCRAM questionnaire contains three 5-item scales measuring sleep quality, diurnal preference, and mood. All items are measured on a 6-point Likert-type scale ranging from 1 (Strongly Disagree) to 6 (Strongly Agree).

CONTACTS AND LOCATIONS:
Locations (1):
- USM, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No